CLINICAL TRIAL: NCT06676683
Title: The Use of Statin in Diabetic Patients Not Known to Have Atherosclerotic Cardiovascular Disease in a Low Income Community
Brief Title: The Use of Statin in Diabetic Patients Not Known to Have Atherosclerotic Cardiovascular Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Islam Abd El-aziz Hassan Mahmoud, Doctor, Sohag University
Other Study IDs: Statin in diabetic patient
Record Dates: First submitted 2024-11-01; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Diabete Type 2
Keywords: Statin - diabetic - Atherosclerotic cardiovascular disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Usage of Statin in diabetic patients — The use of statin in diabetic patients not known to have Atherosclerotic cardiovascular disease in a low income community

SUMMARY:
the use of Statin in diabetic patients and its correlation to the guidelines recommendation.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a chronic disease characterized by hyperglycemia due to insulin resistance resulting in vascular complications. It accounts for approximately 75% of all atherosclerosis-related events.

Moreover, 65% of patients with diabetes die from any type of cardiovascular disease or stroke. Currently, lipid-lowering statin therapy is recommended for the primary prevention of atherosclerotic cardiovascular diseases, as well as for secondary prevention in DM patients with established cardiovascular disease.

The cardiovascular effects of statins extend beyond their effects on lipid fractions and include atherosclerotic plaque stabilization, anti-inflammatory effects, inhibition of vascular smooth muscle cell proliferation, inhibition of platelet function, and improved vascular endothelial function.

Diabetes mellitus (DM) increases cardiovascular disease (CVD) incidence and mortality. While guidelines endorse statin use in type 2 DM (T2DM) to mitigate cardiovascular risks and mortality, challenges like statin initiation and prompt treatment adjustments affect patient outcomes.

According to the ADA and ACC/AHA guidelines, moderate-intensity statin and lifestyle modifcations are recommended for all diabetic patients aged 40-75 without contraindication to statin therapy to achieve an LDL goal of less than 100 mg/dL. Furthermore, high-intensity statin therapy is recommended for patients with cardiovascular risk factors or overt cardiovascular disease to achieve the LDL goal of less than 70 mg/day.

Even though statins should be prescribed for diabetic patients (> 40) regardless of their LDL laboratory values, monitoring their LDL is needed because some patients may have high LDL values even though they are using statins. It is imperative to consider this because high LDL values build up fatty deposits in the arteries, which reduce blood flow, leading to an increased risk of heart attack.

For primary prevention, moderate-dose statin therapy is recommended for those aged $40 years although high-intensity therapy should be considered in the context of additional ASCVD risk factors. The evidence is strong for people with diabetes aged 40-75 years, an age-group well represented in statin trials showing benefit. Since cardiovascular risk is enhanced in people with diabetes, as noted above, individuals who also have multiple other coronary risk factors have increased risk, equivalent to that of those with ASCVD. Therefore, current guidelines recommend that in people with diabetes who are at higher cardiovascular risk, especially those with one or more ASCVD risk factors, high intensity statin therapy should be prescribed to reduce LDL cholesterol by $50% from baseline and to target an LDL cholesterol of <70 mg/dL (<1.8 mmol/L) Five categories for reasons for statin nonuse were finalized after manual annotation: statin-associated side effects/contraindication, guideline discordant clinician practice, clinical inertia, statin hesitancy, and nonspecific reasons. In addition to side effects attributed to prior statin use, if statins were avoided based on pre-existing comorbidities (such as liver disease) or perceived contraindications (including pregnancy) without a trial or challenge, these reasons were categorized within the side effects/contraindication category. This was done because of low individual frequencies for some of these reasons and to comply with privacy regulations that prevent the reporting of groups with fewer than 10 patients. Clinicians avoiding statin use based on lipid levels was considered guideline-discordant practice, given that statin indications for diabetes are primarily independent of lipid levels. Deferral of statin decisions to future visits despite their indications was considered clinical inertia. Statin hesitancy was noted when patients expressed a preference to avoid statins despite discussion of their indication. Nonspecific documentation was recorded when statin nonuse was documented without additional explanation.

ELIGIBILITY:
Inclusion Criteria:

* All diabetic > 18 years.

Exclusion Criteria:

* Diabetic Patients with known to have Atherosclerotic cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Use of Statin in diabetic patients and its correlation to the guidelines recommendation.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
changes in lipid profile in response to treatment with statin in diabetc patients | 12 Weeks
  Guidelines endorse statin use in Type 2 Diabetes Mellitus (T2DM) to mitigate cardiovascular risks and mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Farmer JA. Diabetic dyslipidemia and atherosclerosis: evidence from clinical trials. Curr Diab Rep. 2008 Feb;8(1):71-7. doi: 10.1007/s11892-008-0013-2. PMID 18367002
- [Background] de Vries FM, Denig P, Pouwels KB, Postma MJ, Hak E. Primary prevention of major cardiovascular and cerebrovascular events with statins in diabetic patients: a meta-analysis. Drugs. 2012 Dec 24;72(18):2365-73. doi: 10.2165/11638240-000000000-00000. PMID 23186103
- [Background] Kurihara O, Thondapu V, Kim HO, Russo M, Sugiyama T, Yamamoto E, Fracassi F, Minami Y, Wang Z, Lee H, Yonetsu T, Jang IK. Comparison of Vascular Response to Statin Therapy in Patients With Versus Without Diabetes Mellitus. Am J Cardiol. 2019 May 15;123(10):1559-1564. doi: 10.1016/j.amjcard.2019.02.020. Epub 2019 Feb 22. PMID 30851939
- [Background] Almeida SO, Budoff M. Effect of statins on atherosclerotic plaque. Trends Cardiovasc Med. 2019 Nov;29(8):451-455. doi: 10.1016/j.tcm.2019.01.001. Epub 2019 Jan 7. PMID 30642643
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Sep 10;140(11):e596-e646. doi: 10.1161/CIR.0000000000000678. Epub 2019 Mar 17. No abstract available. PMID 30879355
- [Background] Addendum. 10. Cardiovascular Disease and Risk Management: Standards of Medical Care in Diabetes-2021. Diabetes Care 2021;44(Suppl. 1):S125-S150. Diabetes Care. 2021 Sep;44(9):2183-2185. doi: 10.2337/dc21-ad09a. Epub 2021 Jun 16. No abstract available. PMID 34135017
- [Background] Ogasawara K, Mashiba S, Hashimoto H, Kojima S, Matsuno S, Takeya M, Uchida K, Yajima J. Low-density lipoprotein (LDL), which includes apolipoprotein A-I (apoAI-LDL) as a novel marker of coronary artery disease. Clin Chim Acta. 2008 Nov;397(1-2):42-7. doi: 10.1016/j.cca.2008.07.014. Epub 2008 Jul 18. PMID 18691566
- [Background] Taylor F, Huffman MD, Macedo AF, Moore TH, Burke M, Davey Smith G, Ward K, Ebrahim S. Statins for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD004816. doi: 10.1002/14651858.CD004816.pub5. PMID 23440795
- [Background] Carter AA, Gomes T, Camacho X, Juurlink DN, Shah BR, Mamdani MM. Risk of incident diabetes among patients treated with statins: population based study. BMJ. 2013 May 23;346:f2610. doi: 10.1136/bmj.f2610. PMID 23704171
- [Background] Jellinger PS, Handelsman Y, Rosenblit PD, Bloomgarden ZT, Fonseca VA, Garber AJ, Grunberger G, Guerin CK, Bell DSH, Mechanick JI, Pessah-Pollack R, Wyne K, Smith D, Brinton EA, Fazio S, Davidson M. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY GUIDELINES FOR MANAGEMENT OF DYSLIPIDEMIA AND PREVENTION OF CARDIOVASCULAR DISEASE. Endocr Pract. 2017 Apr;23(Suppl 2):1-87. doi: 10.4158/EP171764.APPGL. PMID 28437620
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Rodriguez F, Maron DJ, Knowles JW, Virani SS, Lin S, Heidenreich PA. Association Between Intensity of Statin Therapy and Mortality in Patients With Atherosclerotic Cardiovascular Disease. JAMA Cardiol. 2017 Jan 1;2(1):47-54. doi: 10.1001/jamacardio.2016.4052. PMID 27829091